CLINICAL TRIAL: NCT02087904
Title: A Phase 2a Study Evaluating the Safety, Efficacy, and Pharmacodynamic Effects of ABT-981 in Patients With Knee Osteoarthritis
Brief Title: A Study Evaluating the Safety, Efficacy, and Pharmacodynamic Effects of ABT-981 in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-741; 2013-003467-60 (EudraCT Number)
Record Dates: First submitted 2014-03-13; First posted 2014-03-14 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2017-01

CONDITIONS: Knee Osteoarthritis; Medial Compartment Knee Osteoarthritis
Keywords: Osteoarthritis; Synovitis; Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Synovitis; Pain | interventions — lutikizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ABT-981 low dose (Experimental): 25 mg ABT-981 subcutaneous (SC) every 2 weeks (E2W)
  Interventions: Biological: ABT-981
- ABT-981 medium dose (Experimental): 100 mg ABT-981 SC E2W
  Interventions: Biological: ABT-981
- ABT-981 high dose (Experimental): 200 mg ABT-981 SC E2W
  Interventions: Biological: ABT-981
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ABT-981
  Other Names: Lutikizumab
  Arms: ABT-981 high dose; ABT-981 low dose; ABT-981 medium dose
Other: Placebo
  Arms: Placebo

SUMMARY:
A Phase 2a, multicenter, randomized, double-blind, parallel group, placebo-controlled study to evaluate the safety, tolerability, efficacy and pharmacokinetic/pharmacodynamic effect of ABT-981 in patients with symptomatic, radiographic, and inflammatory knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographic knee osteoarthritis with Kellgren-Lawrence Grade 2 or 3
2. Body Mass Index (BMI) 18-34 kg/m2
3. One or more clinical signs and symptoms of active inflammation in the index knee

Exclusion Criteria:

1. History of allergic reaction to any constituents of the study drug, or to any Immunoglobulin G (IgG)-containing product
2. History of anaphylactic reaction to any agent
3. Significant trauma or surgery to the index knee
4. Severe knee malalignment
5. Any uncontrolled medical illness or an unstable treatment or therapy

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Levesque, MD, Study Chair — AbbVie

REFERENCES:
- [Derived] Fleischmann RM, Bliddal H, Blanco FJ, Schnitzer TJ, Peterfy C, Chen S, Wang L, Feng S, Conaghan PG, Berenbaum F, Pelletier JP, Martel-Pelletier J, Vaeterlein O, Kaeley GS, Liu W, Kosloski MP, Levy G, Zhang L, Medema JK, Levesque MC. A Phase II Trial of Lutikizumab, an Anti-Interleukin-1alpha/beta Dual Variable Domain Immunoglobulin, in Knee Osteoarthritis Patients With Synovitis. Arthritis Rheumatol. 2019 Jul;71(7):1056-1069. doi: 10.1002/art.40840. Epub 2019 Jun 7. PMID 30653843

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a screening period (approximately 45 days prior to first study drug dose) and a washout period (5 half-lives of the longest acting analgesic used, or 48 hours, whichever was longer, in which all standard of care analgesic medications were discontinued prior to the first study drug dose).
Groups:
- Placebo: Matching placebo SC E2W
- ABT-981 25 mg: 25 mg ABT-981 SC E2W
- ABT-981 100 mg: 100 mg ABT-981 SC E2W
- ABT-981 200 mg: 200 mg ABT-981 SC E2W
Period: Overall Study
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Started | 85 | 89 | 87 | 89
Completed | 60 | 70 | 65 | 64
Not Completed | 25 | 19 | 22 | 25
Not completed — Did Not Receive Study Drug | 0 | 0 | 2 | 1
Not completed — Adverse Event | 8 | 4 | 4 | 12
Not completed — Lack of Efficacy | 3 | 6 | 3 | 2
Not completed — Other | 6 | 2 | 4 | 4
Not completed — Withdrawal by Subject | 8 | 3 | 7 | 4
Not completed — Lost to Follow-up | 0 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat population: all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg | Total
Number analyzed (Participants) | 85 | 89 | 85 | 88 | 347
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.53 (8.850) | 61.63 (7.546) | 60.21 (8.194) | 59.05 (10.273) | 60.11 (8.792)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 63 | 53 | 57 | 225
  Male | 33 | 26 | 32 | 31 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Scores of the Index Knee at Week 16
Description: The WOMAC was developed to assess pain, stiffness, and physical function in subjects with hip and/or knee osteoarthritis. The WOMAC consists of 24 items divided into 3 subscales: Pain (5 items); Stiffness (2 items); and Physical Function (17 items). Each item is rated on an 11-point (0 to 10) numerical rating scale (NRS). The pain sub-score has a range of 0 (no pain) to 50 (maximum pain). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: Modified Intent to Treat population: all subjects who received at least 1 dose of study drug, Last observation carried forward (LOCF; missing responses were imputed by calculation based on the last non-missing post-baseline component values).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 88
score on a scale | -8.9 [-10.96 to -6.90] | -9.2 [-11.23 to -7.23] | -11.8 [-13.84 to -9.75] | -10.1 [-12.10 to -8.10]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.834, ANCOVA — P-value for test of difference between ABT-981 25 mg dose group and Placebo at each postbaseline time point was from an ANCOVA model with treatment, age, and Kellgren-Lawrence (K-L) grade as the main factors and baseline as a covariate; LS Mean Difference = -0.3, 95% CI 2-sided [-3.13 to 2.53]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.05, ANCOVA — P-value for test of difference between ABT-981 100 mg dose group and Placebo at each postbaseline time point was from an ANCOVA model with treatment, age, and K-L grade as the main factors and baseline as a covariate; LS Mean Difference = -2.9, 95% CI 2-sided [-5.73 to 0.01]
Statistical Analysis 3: Comparison: ABT-981 200 mg; Test type: Superiority; p = 0.415, ANCOVA — P-value for test of difference between ABT-981 200 mg dose group and Placebo at each postbaseline time point was from an ANCOVA model with treatment, age, and K-L grade as the main factors and baseline as a covariate; LS Mean Difference = -1.2, 95% CI 2-sided [-4.00 to 1.66]

2. Primary Outcome: Change From Baseline in Quantitative Synovitis of the Index Knee at Week 26
Description: Change in synovitis of the index knee was evaluated using quantitative magnetic resonance imaging (MRI) measurements. MRI quantitative synovitis of the index knee was defined by mean synovial membrane thickness.
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 59 | 65 | 59 | 63
mm | -0.05 [-0.107 to 0.011] | 0.01 [-0.045 to 0.068] | -0.08 [-0.134 to -0.016] | 0.01 [-0.047 to 0.067]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.145, ANCOVA — P-value for test of difference between ABT-981 25 mg dose group and Placebo at each postbaseline time point was from an ANCOVA model with treatment, age, and K-L grade as the main factors and baseline as a covariate; LS Mean Difference = 0.06, 95% CI 2-sided [-0.021 to 0.141]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.52, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.03, 95% CI 2-sided [-0.11 to 0.056]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.159, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0.06, 95% CI 2-sided [-0.023 to 0.139]

3. Primary Outcome: Change From Baseline in Effusion Volume of the Index Knee at Week 26
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 60 | 69 | 67 | 68
mL | 0.03 [-2.498 to 2.562] | 0.26 [-2.113 to 2.624] | -1.04 [-3.421 to 1.347] | -1.49 [-3.868 to 0.898]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.897, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.22, 95% CI 2-sided [-3.193 to 3.642]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.542, ANCOVA — P-value for test of difference between ABT-981 100 dose group and Placebo at each post-baseline time point was from an ANCOVA model with treatment, age, and K-L grade as the main factors and baseline as a covariate; LS Mean Difference = -1.07, 95% CI 2-sided [-4.515 to 2.377]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.385, ANCOVA — P-value for test of difference between ABT-981 200 dose group and Placebo at each post-baseline time point was from an ANCOVA model with treatment, age, and K-L grade as the main factors and baseline as a covariate; LS Mean Difference = -1.52, 95% CI 2-sided [-4.95 to 1.916]

4. Primary Outcome: Change From Baseline in Whole-Organ Magnetic Resonance Imaging Score (WORMS) Semi-Quantitative Synovitis/Effusion Score of the Index Knee at Week 26
Description: Semi-quantitative synovitis/effusion volume WORMS scores were scored as normal (0), < 33% of maximum estimated distention (1), 33% - 66% of maximum estimated distention (2), or > 66% of maximum estimated distention (3).
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 70 | 76 | 70 | 75
score on a scale | 0.07 [-0.057 to 0.193] | -0.01 [-0.130 to 0.113] | -0.08 [-0.205 to 0.043] | -0.07 [-0.196 to 0.048]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.384, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.08, 95% CI 2-sided [-0.249 to 0.096]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.095, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.15, 95% CI 2-sided [-0.324 to 0.026]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.106, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.14, 95% CI 2-sided [-0.314 to 0.03]

5. Secondary Outcome: Change From Baseline in WOMAC Physical Function Scores of the Index Knee at Week 16
Description: The WOMAC was developed to assess pain, stiffness, and physical function in subjects with hip and/or knee osteoarthritis. The WOMAC consists of 24 items divided into 3 subscales: Pain (5 items); Stiffness (2 items); and Physical Function (17 items). Each item is rated on an 11-point (0 to 10) NRS. The WOMAC physical function subscale score was 0 (normal) to 170 (least physical function). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: Modified intent to Treat population: all participants who received at least 1 dose of study drug, LOCF (missing responses were imputed by calculation based on the last non-missing post-baseline component values).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 87
score on a scale | -28.7 [-35.30 to -22.15] | -29.8 [-36.27 to -23.32] | -36.3 [-42.90 to -29.69] | -32.1 [-38.64 to -25.63]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.818, ANCOVA — P-value for test of difference between ABT-981 25 mg dose group and placebo at each postbaseline time point is from an ANCOVA model with treatment, age, K-L grade as the main factors and baseline as a covariate; LS Mean Difference = -1.1, 95% CI 2-sided [-10.22 to 8.08]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.109, ANCOVA — P-value for test of difference between ABT-981 100 mg dose group and placebo at each postbaseline time point is from an ANCOVA model with treatment, age, K-L grade as the main factors and baseline as a covariate; LS Mean Difference = -7.6, 95% CI 2-sided [-16.83 to 1.69]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.465, ANCOVA — P-value for test of difference between ABT-981 200 mg dose group and placebo at each postbaseline time point is from an ANCOVA model with treatment, age, K-L grade as the main factors and baseline as a covariate; LS Mean Difference = -3.4, 95% CI 2-sided [-12.58 to 5.76]

6. Secondary Outcome: Change From Baseline in WOMAC Physical Function Scores of the Index Knee at Week 26
Description: as for outcome 5
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 87
score on a scale | -29.7 [-36.61 to -22.75] | -31.8 [-38.62 to -24.98] | -38.9 [-45.83 to -31.92] | -36.9 [-43.71 to -30.00]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.666, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-11.76 to 7.52]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.065, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LS Mean Difference = -9.2, 95% CI 2-sided [-18.95 to 0.56]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.145, ANCOVA — [p-value comment as in outcome 5, analysis 3]; LS Mean Difference = -7.2, 95% CI 2-sided [-16.84 to 2.49]

7. Secondary Outcome: Change From Baseline in WOMAC Physical Function Scores of the Index Knee at Week 52
Description: as for outcome 5
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 87
score on a scale | -32.9 [-40.66 to -25.12] | -36.1 [-43.76 to -28.46] | -38.7 [-46.52 to -30.92] | -39.7 [-47.37 to -32.00]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.558, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -3.2, 95% CI 2-sided [-14.03 to 7.59]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.295, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LS Mean Difference = -5.8, 95% CI 2-sided [-16.77 to 5.11]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.218, ANCOVA — [p-value comment as in outcome 5, analysis 3]; LS Mean Difference = -6.8, 95% CI 2-sided [-17.63 to 4.04]

8. Secondary Outcome: Change From Baseline in WOMAC Pain Scores of the Index Knee at Week 26
Description: as for outcome 1
Time Frame: Baseline, Week 26
Population: Modified intent to Treat population: all subjects who received at least 1 dose of study drug, LOCF (missing responses were imputed by calculation based on the last non-missing post-baseline component values).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 88
score on a scale | -9.2 [-11.29 to -7.07] | -9.8 [-11.90 to -7.75] | -11.9 [-13.99 to -9.76] | -11.6 [-13.65 to -9.51]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.664, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-3.58 to 2.28]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.075, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LS Mean Difference = -2.7, 95% CI 2-sided [-5.67 to 0.28]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.107, ANCOVA — [p-value comment as in outcome 5, analysis 3]; LS Mean Difference = -2.4, 95% CI 2-sided [-5.33 to 0.52]

9. Secondary Outcome: Change From Baseline in WOMAC Pain Scores of the Index Knee at Week 52
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 88
score on a scale | -10.0 [-12.24 to -7.68] | -11.0 [-13.29 to -8.80] | -12.1 [-14.42 to -9.84] | -12.2 [-14.49 to -10.0]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.5, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 0.5, 95% CI 2-sided [-4.26 to 2.08]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.186, ANCOVA — [p-value comment as in outcome 5, analysis 2]; LS Mean Difference = -2.2, 95% CI 2-sided [-5.39 to 1.05]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.157, ANCOVA — [p-value comment as in outcome 5, analysis 3]; LS Mean Difference = -2.3, 95% CI 2-sided [-5.46 to 0.88]

10. Secondary Outcome: Change From Baseline in Global Total Bone Marrow Lesion (BML) Score of the Index Knee Magnetic Resonance Imaging (MRI) at Week 26
Description: BMLs in 15 regions were measured with MRI, and graded as 0 (normal), 1 (mild; < 25% of region), 2 (moderate; 25% - 50% of region), or 3 (severe; > 50% of region). The global total BML score was the sum of the 15 component scores, and ranged from 0 (normal) to 45 (severe).
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 69 | 76 | 69 | 75
score on a scale | 0.1 [-0.24 to 0.43] | 0.3 [0.01 to 0.65] | -0.0 [-0.37 to 0.29] | 0.1 [-0.22 to 0.43]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.319, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.23 to 0.69]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.564, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.33]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.966, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0, 95% CI 2-sided [-0.45 to 0.47]

11. Secondary Outcome: Change From Baseline in Global Total BML Score of the Index Knee MRI at Week 52
Description: as for outcome 10
Time Frame: Baseline, Week 52
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 56 | 66 | 61 | 66
score on a scale | 0.1 [-0.34 to 0.48] | 0.2 [-0.16 to 0.60] | 0.1 [-0.30 to 0.48] | 0.0 [-0.36 to 0.39]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.602, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.41 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.953, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0, 95% CI 2-sided [-0.55 to 0.58]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.83, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.61 to 0.49]

12. Secondary Outcome: Change From Baseline in Index Knee Intermittent and Constant Osteoarthritis Pain (ICOAP) Scores at Week 16
Description: The ICOAP is a multidimensional osteoarthritis-specific measure designed to comprehensively evaluate the pain experience in patients with hip or knee osteoarthritis. The ICOAP includes 11 items (5 constant pain items; 6 intermittent pain items). Each item is rated on a 0 to 4 point scale with a 7-day recall period. The raw maximum intermittent pain score ranges from 0 to 24, transformed to a reported scale of 0 (no pain) to 100 (worst pain). The raw maximum constant pain score ranges from 0 to 20, transformed to a reported scale of 0 (no pain) to 100 (worst pain).
Time Frame: Baseline, Week 16
Population: Modified Intent to Treat population: all subjects who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 75 | 84 | 76 | 77
score on a scale
  Intermittent Pain | -20.2 [-24.32 to -16.08] | -19.5 [-23.40 to -15.58] | -21.3 [-25.40 to -17.26] | -18.8 [-22.92 to -14.71]
  Constant Pain | -18.6 [-22.88 to -14.33] | -17.7 [-21.73 to -13.62] | -24.2 [-28.39 to -19.94] | -20.0 [-24.24 to -15.72]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Intermittent pain; Test type: Superiority; p = 0.804, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.7, 95% CI 2-sided [-4.91 to 6.33]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Intermittent pain; Test type: Superiority; p = 0.699, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -1.1, 95% CI 2-sided [-6.9 to 4.63]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Intermittent pain; Test type: Superiority; p = 0.636, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 1.4, 95% CI 2-sided [-4.37 to 7.14]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Constant pain; Test type: Superiority; p = 0.756, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.9, 95% CI 2-sided [-4.91 to 6.76]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Constant pain; Test type: Superiority; p = 0.068, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -5.6, 95% CI 2-sided [-11.55 to 0.42]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Constant pain; Test type: Superiority; p = 0.649, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -1.4, 95% CI 2-sided [-7.34 to 4.58]

13. Secondary Outcome: Change From Baseline in Index Knee ICOAP Scores at Week 26
Description: as for outcome 12
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all subjects who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 68 | 75 | 72 | 73
score on a scale
  Intermittent Pain | -18.7 [-23.21 to -14.21] | -19.7 [-23.99 to -15.42] | -21.3 [-25.66 to -16.98] | -21.7 [-26.11 to -17.38]
  Constant Pain | -19.6 [-24.22 to -14.96] | -18.8 [-23.26 to -14.42] | -21.6 [-26.05 to -17.08] | -22.1 [-26.61 to -17.61]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Intermittent pain; Test type: Superiority; p = 0.75, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -1, 95% CI 2-sided [-7.14 to 5.14]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Intermittent pain; Test type: Superiority; p = 0.409, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2.6, 95% CI 2-sided [-8.82 to 3.6]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Intermittent pain; Test type: Superiority; p = 0.338, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -3, 95% CI 2-sided [-9.24 to 3.18]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Constant pain; Test type: Superiority; p = 0.817, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.7, 95% CI 2-sided [-5.59 to 7.08]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Constant pain; Test type: Superiority; p = 0.544, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -2, 95% CI 2-sided [-8.37 to 4.43]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Constant pain; Test type: Superiority; p = 0.437, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -2.5, 95% CI 2-sided [-8.91 to 3.86]

14. Secondary Outcome: Change From Baseline in Index Knee ICOAP Scores at Week 52
Description: as for outcome 12
Time Frame: Baseline, Week 52
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 58 | 70 | 66 | 66
score on a scale
  Intermittent Pain | -23.2 [-28.51 to -17.83] | -25.4 [-30.21 to -20.51] | -23.6 [-28.53 to -18.64] | -27.2 [-32.19 to -22.14]
  Constant Pain | -20.6 [-25.93 to -15.21] | -21.8 [-26.70 to -16.94] | -25.2 [-30.14 to -20.17] | -29.7 [-34.78 to -24.66]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Intermittent pain; Test type: Superiority; p = 0.545, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -2.2, 95% CI 2-sided [-9.31 to 4.92]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Intermittent pain; Test type: Superiority; p = 0.909, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.4, 95% CI 2-sided [-7.65 to 6.81]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Intermittent pain; Test type: Superiority; p = 0.278, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -4.0, 95% CI 2-sided [-11.23 to 3.25]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Constant pain; Test type: Superiority; p = 0.732, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-8.42 to 5.92]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Constant pain; Test type: Superiority; p = 0.216, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -4.6, 95% CI 2-sided [-11.86 to 2.69]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Constant pain; Test type: Superiority; p = 0.014, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -9.2, 95% CI 2-sided [-16.42 to -1.88]

15. Secondary Outcome: Change From Baseline In Index Knee Pain Intensity at Week 16
Description: The index knee pain intensity was assessed in 3 different ways using an 11 -point NRS (0 to 10 points representing 'no pain' to 'worst possible pain'). Subjects were asked to enter: 1) average pain intensity during the past week (7-day recall period); 2) the worst pain during activity over the past 24 hours; 3) pain intensity before and after a 40 meter walk (performance pain, before and after). The 40 meter fast paced walk test is a test of short distance walking activity, walking speed over short distances and changing direction during walking. Individuals taking the test should walk as quickly but as safely as possible, without running, along a walkway and then turn around, and repeat again for a total distance of 40 m (132 feet). The total time taken to walk the 40 meters is recorded.
Time Frame: Baseline, Week 16
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 75 | 84 | 77 | 77
units on a scale
  7-Day Recall Period | -2.4 [-2.86 to -1.97] | -2.4 [-2.79 to -1.95] | -2.7 [-3.09 to -2.22] | -2.1 [-2.55 to -1.67]
  Activity Pain | -2.3 [-2.85 to -1.82] | -2.4 [-2.85 to -1.87] | -2.7 [-3.19 to -2.17] | -2.1 [-2.59 to -1.56]
  Performance Pain (Before) | -2.4 [-2.82 to -1.89] | -2.1 [-2.58 to -1.70] | -2.5 [-2.97 to -2.06] | -2.1 [-2.52 to -1.60]
  Performance Pain (After) | -2.6 [-3.07 to -2.11] | -2.4 [-2.90 to -2.00] | -2.7 [-3.16 to -2.22] | -2.3 [-2.77 to -1.82]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; 7-day recall period; Test type: Superiority; p = 0.874, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.56 to 0.66]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; 7-day recall period; Test type: Superiority; p = 0.451, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.86 to 0.38]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; 7-day recall period; Test type: Superiority; p = 0.331, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.31 to 0.93]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Activity pain; Test type: Superiority; p = 0.932, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.73 to 0.67]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Activity pain; Test type: Superiority; p = 0.344, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.3, 95% CI 2-sided [-1.07 to 0.37]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Activity pain; Test type: Superiority; p = 0.489, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.47 to 0.97]
Statistical Analysis 7: Comparison: Placebo vs ABT-981 25 mg; Performance pain (before); Test type: Superiority; p = 0.498, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.42 to 0.85]
Statistical Analysis 8: Comparison: Placebo vs ABT-981 100 mg; Performance pain (before); Test type: Superiority; p = 0.637, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.8 to 0.49]
Statistical Analysis 9: Comparison: Placebo vs ABT-981 200 mg; Performance pain (before); Test type: Superiority; p = 0.367, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.35 to 0.94]
Statistical Analysis 10: Comparison: Placebo vs ABT-981 25 mg; Performance pain (after); Test type: Superiority; p = 0.67, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.51 to 0.79]
Statistical Analysis 11: Comparison: Placebo vs ABT-981 100 mg; Performance pain (after); Test type: Superiority; p = 0.776, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.76 to 0.57]
Statistical Analysis 12: Comparison: Placebo vs ABT-981 200 mg; Performance pain (after); Test type: Superiority; p = 0.387, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.37 to 0.96]

16. Secondary Outcome: Change From Baseline In Index Knee Pain Intensity at Week 26
Description: as for outcome 15
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 68 | 75 | 73 | 73
units on a scale
  7-Day Recall Period | -2.2 [-2.76 to -1.73] | -2.4 [-2.89 to -1.91] | -2.8 [-3.29 to -2.31] | -2.5 [-2.98 to -1.99]
  Activity Pain | -2.5 [-3.07 to -1.91] | -2.5 [-3.10 to -1.99] | -2.8 [-3.37 to -2.25] | -2.5 [-3.10 to -1.97]
  Performance Pain (Before) | -2.2 [-2.72 to -1.70] | -2.2 [-2.68 to -1.71] | -2.6 [-3.13 to -2.16] | -2.7 [-3.15 to -2.17]
  Performance Pain (After): number analyzed (Participants) | 67 | 75 | 72 | 73
  Performance Pain (After) | -2.5 [-3.01 to -1.98] | -2.4 [-2.90 to -1.92] | -3.0 [-3.53 to -2.54] | -2.6 [-3.13 to -2.13]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; 7-day recall period; Test type: Superiority; p = 0.661, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.86 to 0.54]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; 7-day recall period; Test type: Superiority; p = 0.122, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.26 to 0.15]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; 7-day recall period; Test type: Superiority; p = 0.507, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.94 to 0.47]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Activity pain; Test type: Superiority; p = 0.892, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.85 to 0.74]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Activity pain; Test type: Superiority; p = 0.433, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.3, 95% CI 2-sided [-1.12 to 0.48]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Activity pain; Test type: Superiority; p = 0.92, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.84 to 0.76]
Statistical Analysis 7: Comparison: Placebo vs ABT-981 25 mg; Performance pain (before); Test type: Superiority; p = 0.957, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.68 to 0.71]
Statistical Analysis 8: Comparison: Placebo vs ABT-981 100 mg; Performance pain (before); Test type: Superiority; p = 0.222, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.13 to 0.26]
Statistical Analysis 9: Comparison: Placebo vs ABT-981 200 mg; Performance pain (before); Test type: Superiority; p = 0.209, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.15 to 0.25]
Statistical Analysis 10: Comparison: Placebo vs ABT-981 25 mg; Performance pain (after); Test type: Superiority; p = 0.813, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.62 to 0.79]
Statistical Analysis 11: Comparison: Placebo vs ABT-981 100 mg; Performance pain (after); Test type: Superiority; p = 0.135, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.25 to 0.17]
Statistical Analysis 12: Comparison: Placebo vs ABT-981 200 mg; Performance pain (after); Test type: Superiority; p = 0.679, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.85 to 0.57]

17. Secondary Outcome: Change From Baseline In Index Knee Pain Intensity at Week 52
Description: as for outcome 15
Time Frame: Baseline, Week 52
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 58 | 70 | 67 | 66
units on a scale
  7-Day Recall Period | -2.9 [-3.51 to -2.35] | -2.9 [-3.45 to -2.39] | -2.9 [-3.43 to -2.35] | -3.1 [-3.65 to -2.56]
  Activity Pain | -2.8 [-3.48 to -2.16] | -3.0 [-3.64 to -2.43] | -3.2 [-3.77 to -2.55] | -3.0 [-3.65 to -2.40]
  Performance Pain (Before) | -2.6 [-3.14 to -2.03] | -2.7 [-3.24 to -2.23] | -3.0 [-3.51 to -2.49] | -2.9 [-3.46 to -2.41]
  Performance Pain (After) | -2.9 [-3.47 to -2.33] | -3.0 [-3.53 to -2.50] | -3.4 [-3.90 to -2.86] | -3.2 [-3.69 to -2.62]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; 7-day recall period; Test type: Superiority; p = 0.978, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.76 to 0.79]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; 7-day recall period; Test type: Superiority; p = 0.925, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.75 to 0.82]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; 7-day recall period; Test type: Superiority; p = 0.659, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.96 to 0.61]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Activity pain; Test type: Superiority; p = 0.633, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.1 to 0.67]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Activity pain; Test type: Superiority; p = 0.46, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.3, 95% CI 2-sided [-1.23 to 0.56]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Activity pain; Test type: Superiority; p = 0.663, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.1 to 0.7]
Statistical Analysis 7: Comparison: Placebo vs ABT-981 25 mg; Performance pain (before); Test type: Superiority; p = 0.696, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.89 to 0.59]
Statistical Analysis 8: Comparison: Placebo vs ABT-981 100 mg; Performance pain (before); Test type: Superiority; p = 0.278, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.16 to 0.34]
Statistical Analysis 9: Comparison: Placebo vs ABT-981 200 mg; Performance pain (before); Test type: Superiority; p = 0.357, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.1 to 0.4]
Statistical Analysis 10: Comparison: Placebo vs ABT-981 25 mg; Performance pain (after); Test type: Superiority; p = 0.761, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.87 to 0.64]
Statistical Analysis 11: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.218, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.02 to 0.51]
Statistical Analysis 12: Comparison: Placebo vs ABT-981 200 mg; Performance pain (after); Test type: Superiority; p = 0.513, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.3, 95% CI 2-sided [-1.02 to 0.51]

18. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Arthritis of the Index Knee at Week 16
Description: The PGA is a single item for evaluating overall osteoarthritis disease activity. PGA is assessed using an 11-point NRS of 0 to 10 points (representing best to worst disease status, respectively), with a 7-day recall period.
Time Frame: Baseline, Week 16
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 75 | 84 | 77 | 77
units on a scale | -2.5 [-2.94 to -2.01] | -2.4 [-2.80 to -1.92] | -2.9 [-3.34 to -2.42] | -2.6 [-3.08 to -2.15]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.728, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.52 to 0.75]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.219, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.06 to 0.24]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.673, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.79 to 0.51]

19. Secondary Outcome: Change From Baseline in PGA of Arthritis of the Index Knee at Week 26
Description: as for outcome 18
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 68 | 75 | 73 | 73
units on a scale | -2.4 [-2.96 to -1.91] | -2.4 [-2.94 to -1.94] | -3.0 [-3.48 to -2.47] | -2.7 [-3.18 to -2.16]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.984, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.73 to 0.71]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.145, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.26 to 0.19]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.527, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.96 to 0.49]

20. Secondary Outcome: Change From Baseline in PGA of Arthritis of the Index Knee at Week 52
Description: as for outcome 18
Time Frame: Baseline, Week 52
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 58 | 70 | 67 | 66
units on a scale | -3.0 [-3.62 to -2.44] | -2.9 [-3.48 to -2.41] | -3.2 [-3.71 to -2.62] | -3.5 [-4.01 to -2.89]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.836, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.71 to 0.87]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.738, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.94 to 0.66]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.3, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.22 to 0.38]

21. Secondary Outcome: Change From Baseline in Cartilage Volume of the Index Knee at Week 26
Description: Cartilage volume of the global knee, the medial central condyle + plateau, and the medial condyle + plateau was measured using MRI.
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm^3
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 58 | 65 | 53 | 66
mm^3
  Global Knee | -326.0 [-400.83 to -251.13] | -325.5 [-397.10 to -253.83] | -322.4 [-400.20 to -244.61] | -359.0 [-429.72 to -288.35]
  Medial Central Condyle + Plateau | -59.1 [-83.12 to -35.10] | -54.9 [-77.83 to -31.90] | -50.1 [-75.13 to -25.07] | -57.5 [-80.12 to -34.88]
  Medial Condyle + Plateau | -128.6 [-166.76 to -90.50] | -126.5 [-163.03 to -90.02] | -124.5 [-164.13 to -84.86] | -114.9 [-150.86 to -78.90]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Global knee; Test type: Superiority; p = 0.992, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.5, 95% CI 2-sided [-101.59 to 102.62]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Global knee; Test type: Superiority; p = 0.948, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 3.6, 95% CI 2-sided [-103.95 to 111.10]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Global knee; Test type: Superiority; p = 0.523, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -33.1, 95% CI 2-sided [-134.76 to 68.65]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.799, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 4.2, 95% CI 2-sided [-28.47 to 36.95]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.609, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 9.0, 95% CI 2-sided [-25.62 to 43.64]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.923, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 1.6, 95% CI 2-sided [-30.97 to 34.19]
Statistical Analysis 7: Comparison: Placebo vs ABT-981 25 mg; Medial condyle + plateau; Test type: Superiority; p = 0.937, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 2.1, 95% CI 2-sided [-49.88 to 54.08]
Statistical Analysis 8: Comparison: Placebo vs ABT-981 100 mg; Medial condyle + plateau; Test type: Superiority; p = 0.882, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 4.1, 95% CI 2-sided [-50.68 to 58.95]
Statistical Analysis 9: Comparison: Placebo vs ABT-981 200 mg; Medial condyle + plateau; Test type: Superiority; p = 0.602, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 13.8, 95% CI 2-sided [-38.05 to 65.55]

22. Secondary Outcome: Change From Baseline in Cartilage Volume of the Index Knee at Week 52
Description: as for outcome 21
Time Frame: Baseline, Week 52
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm^3
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 49 | 57 | 50 | 56
mm^3
  Global Knee | -557.0 [-659.86 to -454.10] | -598.7 [-694.66 to -502.76] | -554.3 [-654.92 to -453.60] | -583.1 [-678.88 to -487.23]
  Medial Central Condyle + Plateau | -101.2 [-134.56 to -67.79] | -126.3 [-157.5 to -95.09] | -90.1 [-122.89 to -57.29] | -113.0 [-144.08 to -81.84]
  Medial Condyle + Plateau | -214.7 [-273.77 to -155.64] | -255.0 [-310.03 to -199.97] | -190.3 [-248.05 to -132.51] | -242.8 [-297.71 to -187.86]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Global knee; Test type: Superiority; p = 0.554, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -41.7, 95% CI 2-sided [-180.49 to 97.04]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Global knee; Test type: Superiority; p = 0.97, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 2.7, 95% CI 2-sided [-140.86 to 146.31]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Global knee; Test type: Superiority; p = 0.713, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -26.1, 95% CI 2-sided [-165.47 to 113.32]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.272, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -25.1, 95% CI 2-sided [-70.12 to 19.88]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.64, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 11.1, 95% CI 2-sided [-35.63 to 57.8]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.608, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -11.8, 95% CI 2-sided [-56.94 to 33.38]
Statistical Analysis 7: Comparison: Placebo vs ABT-981 25 mg; Medial condyle + plateau; Test type: Superiority; p = 0.319, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -40.3, 95% CI 2-sided [-119.88 to 39.3]
Statistical Analysis 8: Comparison: Placebo vs ABT-981 100 mg; Medial condyle + plateau; Test type: Superiority; p = 0.56, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 24.4, 95% CI 2-sided [-58.05 to 106.91]
Statistical Analysis 9: Comparison: Placebo vs ABT-981 200 mg; Medial condyle + plateau; Test type: Superiority; p = 0.489, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -28.1, 95% CI 2-sided [-107.97 to 51.82]

23. Secondary Outcome: Change From Baseline in Cartilage Thickness of the Index Knee at Week 26
Description: Cartilage thickness of the global knee, the medial central condyle + plateau, and the medial condyle + plateau was measured using MRI.
Time Frame: Baseline, Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 58 | 65 | 53 | 66
mm
  Global Knee | -0.047 [-0.058 to -0.036] | -0.047 [-0.058 to -0.037] | -0.048 [-0.059 to -0.037] | -0.052 [-0.062 to -0.041]
  Medial Central Condyle + Plateau | -0.085 [-0.122 to -0.048] | -0.077 [-0.113 to -0.042] | -0.074 [-0.113 to -0.036] | -0.076 [-0.111 to -0.041]
  Medial Condyle + Plateau | -0.046 [-0.060 to -0.031] | -0.045 [-0.059 to -0.031] | -0.047 [-0.062 to -0.032] | -0.044 [-0.058 to -0.031]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Global knee; Test type: Superiority; p = 0.972, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.015 to 0.015]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Global knee; Test type: Superiority; p = 0.929, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.001, 95% CI 2-sided [-0.017 to 0.015]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Global knee; Test type: Superiority; p = 0.543, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.005, 95% CI 2-sided [-0.02 to 0.01]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.752, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.008, 95% CI 2-sided [-0.043 to 0.059]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.691, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.011, 95% CI 2-sided [-0.042 to 0.064]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.71, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0.01, 95% CI 2-sided [-0.041 to 0.06]
Statistical Analysis 7: Comparison: Placebo vs ABT-981 25 mg; Medial condyle + plateau; Test type: Superiority; p = 0.965, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-0.019 to 0.02]
Statistical Analysis 8: Comparison: Placebo vs ABT-981 100 mg; Medial condyle + plateau; Test type: Superiority; p = 0.885, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.002, 95% CI 2-sided [-0.022 to 0.019]
Statistical Analysis 9: Comparison: Placebo vs ABT-981 200 mg; Medial condyle + plateau; Test type: Superiority; p = 0.887, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = 0.001, 95% CI 2-sided [-0.018 to 0.021]

24. Secondary Outcome: Change From Baseline in Cartilage Thickness of the Index Knee at Week 52
Description: as for outcome 23
Time Frame: Baseline, Week 52
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, observed cases.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 49 | 57 | 50 | 56
mm
  Global Knee | -0.081 [-0.095 to -0.066] | -0.085 [-0.099 to -0.072] | -0.081 [-0.095 to -0.067] | -0.083 [-0.097 to -0.070]
  Medial Central Condyle + Plateau | -0.136 [-0.187 to -0.084] | -0.176 [-0.224 to -0.127] | -0.113 [-0.163 to -0.062] | -0.141 [-0.190 to -0.093]
  Medial Condyle + Plateau | -0.084 [-0.106 to -0.063] | -0.096 [-0.117 to -0.076] | -0.073 [-0.094 to -0.052] | -0.087 [-0.107 to -0.067]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Global knee; Test type: Superiority; p = 0.619, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.005, 95% CI 2-sided [-0.024 to 0.014]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Global knee; Test type: Superiority; p = 0.952, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.001, 95% CI 2-sided [-0.02 to 0.019]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Global knee; Test type: Superiority; p = 0.765, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.003, 95% CI 2-sided [-0.022 to 0.016]
Statistical Analysis 4: Comparison: Placebo vs ABT-981 25 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.258, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.04, 95% CI 2-sided [-0.11 to 0.03]
Statistical Analysis 5: Comparison: Placebo vs ABT-981 100 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.535, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.023, 95% CI 2-sided [-0.049 to 0.094]
Statistical Analysis 6: Comparison: Placebo vs ABT-981 200 mg; Medial central condyle + plateau; Test type: Superiority; p = 0.866, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.006, 95% CI 2-sided [-0.076 to 0.064]
Statistical Analysis 7: Comparison: Placebo vs ABT-981 25 mg; Medial condyle + plateau; Test type: Superiority; p = 0.413, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.012, 95% CI 2-sided [-0.041 to 0.017]
Statistical Analysis 8: Comparison: Placebo vs ABT-981 100 mg; Medial condyle + plateau; Test type: Superiority; p = 0.445, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = 0.012, 95% CI 2-sided [-0.018 to 0.042]
Statistical Analysis 9: Comparison: Placebo vs ABT-981 200 mg; Medial condyle + plateau; Test type: Superiority; p = 0.835, ANCOVA — [p-value comment as in outcome 1, analysis 3]; LS Mean Difference = -0.003, 95% CI 2-sided [-0.032 to 0.026]

25. Secondary Outcome: Outcome Measures in Rheumatology Clinical Trials/Osteoarthritis Research Society International (OMERACT/OARSI) Response Rate at Week 16
Description: Percentage of participants classified as OMERACT-OARSI responders at Week 16. A subject was considered an OMERACT-OARSI responder if any of the following 3 criteria were met: 1. WOMAC Pain (in 0 - 100 scale) improvement ≥ 50% and absolute reduction ≥ 20 as compared to the baseline; or 2. WOMAC Function (in normalized 0 - 100 scale) improvement ≥ 50% and absolute reduction ≥ 20 as compared to the baseline; or 3. At least 2 of the following 3 are met: WOMAC Pain improvement ≥ 20% and absolute reduction (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline; WOMAC Function improvement ≥ 20% and absolute reduction (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline; PGA improvement ≥ 20% and absolute change (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline. Response rate 95% confidence interval based on normal approximation.
Time Frame: Week 16
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 87
percentage of participants | 60.0 [49.6 to 70.4] | 67.0 [57.2 to 76.9] | 72.6 [63.1 to 82.2] | 65.5 [55.5 to 75.5]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.311, Cochran-Mantel-Haenszel — P-value for test of difference between each ABT-981 dose group and Placebo was from a Cochran-Mantel-Haenszel test using age group and K-L grade as stratification factors; Response Rate Difference = 7.0, 95% CI 2-sided [-7.3 to 21.4]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.435, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Response Rate Difference = 5.5, 95% CI 2-sided [-8.9 to 19.9]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.435, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Response Rate Difference = 5.5, 95% CI 2-sided [-8.9 to 19.9]

26. Secondary Outcome: Outcome Measures in Rheumatology Clinical Trials/Osteoarthritis Research Society International (OMERACT/OARSI) Response Rate at Week 26
Description: Percentage of participants classified as OMERACT-OARSI responders at Week 26. A subject was considered an OMERACT-OARSI responder if any of the following 3 criteria were met: 1. WOMAC Pain (in 0 - 100 scale) improvement ≥ 50% and absolute reduction ≥ 20 as compared to the baseline; or 2. WOMAC Function (in normalized 0 - 100 scale) improvement ≥ 50% and absolute reduction ≥ 20 as compared to the baseline; or 3. At least 2 of the following 3 are met: WOMAC Pain improvement ≥ 20% and absolute reduction (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline; WOMAC Function improvement ≥ 20% and absolute reduction (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline; PGA improvement ≥ 20% and absolute change (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline. Response rate 95% confidence interval based on normal approximation.
Time Frame: Week 26
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 88
percentage of participants | 62.4 [52.1 to 72.7] | 64.8 [54.8 to 74.8] | 66.7 [56.6 to 76.7] | 72.7 [63.4 to 82.0]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.744, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Response Rate Difference = 2.4, 95% CI 2-sided [-11.9 to 16.8]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.581, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Response Rate Difference = 4.3, 95% CI 2-sided [-10.1 to 18.7]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.146, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Response Rate Difference = 10.4, 95% CI 2-sided [-3.5 to 24.3]

27. Secondary Outcome: Outcome Measures in Rheumatology Clinical Trials/Osteoarthritis Research Society International (OMERACT/OARSI) Response Rate at Week 52
Description: Percentage of participants classified as OMERACT-OARSI responders at Week 52. A subject was considered an OMERACT-OARSI responder if any of the following 3 criteria were met: 1. WOMAC Pain (in 0 - 100 scale) improvement ≥ 50% and absolute reduction ≥ 20 as compared to the baseline; or 2. WOMAC Function (in normalized 0 - 100 scale) improvement ≥ 50% and absolute reduction ≥ 20 as compared to the baseline; or 3. At least 2 of the following 3 are met: WOMAC Pain improvement ≥ 20% and absolute reduction (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline; WOMAC Function improvement ≥ 20% and absolute reduction (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline; PGA improvement ≥ 20% and absolute change (in normalized 0 - 100 scale) ≥ 10 as compared to the baseline. Response rate 95% confidence interval based on normal approximation.
Time Frame: Week 52
Population: Modified Intent to Treat population: all participants who received at least 1 dose of study drug, LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Number analyzed (Participants) | 85 | 88 | 84 | 88
percentage of participants | 70.6 [60.9 to 80.3] | 69.3 [59.7 to 79.0] | 71.4 [61.8 to 81.1] | 72.7 [63.4 to 82.0]
Statistical Analysis 1: Comparison: Placebo vs ABT-981 25 mg; Test type: Superiority; p = 0.824, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Response Rate Difference = -1.3, 95% CI 2-sided [-14.9 to 12.4]
Statistical Analysis 2: Comparison: Placebo vs ABT-981 100 mg; Test type: Superiority; p = 0.964, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Response Rate Difference = 0.8, 95% CI 2-sided [-12.8 to 14.5]
Statistical Analysis 3: Comparison: Placebo vs ABT-981 200 mg; Test type: Superiority; p = 0.763, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Response Rate Difference = 2.1, 95% CI 2-sided [-11.3 to 15.6]

ADVERSE EVENTS:
Time Frame: up to Week 52 (or last dose of study drug) plus 70 days
Description: Safety population: all participants who took at least one dose of study drug.
Arm/Group | Placebo | ABT-981 25 mg | ABT-981 100 mg | ABT-981 200 mg
Serious Adverse Events (participants affected / at risk) | 8/85 | 11/89 | 8/85 | 4/88
Other Adverse Events (participants affected / at risk) | 66/85 | 63/89 | 65/85 | 75/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | ABT-981 25 mg (N=89) | ABT-981 100 mg (N=85) | ABT-981 200 mg (N=88)
ADRENAL HAEMORRHAGE (Endocrine disorders) | 0 | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 1 | 0
LIVER DISORDER (Hepatobiliary disorders) | 1 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0 | 0 | 0
PERITONITIS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
PROCEDURAL INTESTINAL PERFORATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
AQUEDUCTAL STENOSIS (Nervous system disorders) | 0 | 0 | 1 | 0
BRAIN OEDEMA (Nervous system disorders) | 0 | 0 | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0 | 0
HYDROCEPHALUS (Nervous system disorders) | 0 | 0 | 1 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 0 | 1 | 0
SEIZURE (Nervous system disorders) | 0 | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 0
ALVEOLITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | ABT-981 25 mg (N=89) | ABT-981 100 mg (N=85) | ABT-981 200 mg (N=88)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 12 | 12 | 21
DIARRHOEA (Gastrointestinal disorders) | 7 | 6 | 5 | 9
NAUSEA (Gastrointestinal disorders) | 3 | 4 | 6 | 6
FATIGUE (General disorders) | 12 | 4 | 5 | 7
INJECTION SITE ERYTHEMA (General disorders) | 1 | 4 | 7 | 5
INJECTION SITE PAIN (General disorders) | 7 | 2 | 2 | 1
INJECTION SITE RASH (General disorders) | 3 | 3 | 7 | 8
INJECTION SITE REACTION (General disorders) | 0 | 6 | 8 | 12
PAIN (General disorders) | 6 | 3 | 4 | 4
BRONCHITIS (Infections and infestations) | 2 | 5 | 1 | 4
INFLUENZA (Infections and infestations) | 10 | 2 | 5 | 4
NASOPHARYNGITIS (Infections and infestations) | 16 | 9 | 13 | 17
SINUSITIS (Infections and infestations) | 1 | 5 | 3 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 8 | 7 | 12
URINARY TRACT INFECTION (Infections and infestations) | 4 | 3 | 5 | 8
CONTUSION (Injury, poisoning and procedural complications) | 3 | 9 | 2 | 5
FALL (Injury, poisoning and procedural complications) | 3 | 5 | 3 | 8
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 3 | 6 | 2 | 2
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 3 | 13 | 13
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16 | 16 | 19 | 14
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14 | 8 | 11 | 14
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4 | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 9
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 | 5 | 7 | 5
DIZZINESS (Nervous system disorders) | 1 | 3 | 6 | 3
HEADACHE (Nervous system disorders) | 22 | 14 | 14 | 21
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 5 | 5
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5 | 7
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 6 | 5 | 4
RASH (Skin and subcutaneous tissue disorders) | 3 | 2 | 6 | 4
HYPERTENSION (Vascular disorders) | 6 | 7 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.